CLINICAL TRIAL: NCT04508140
Title: Phase IIa Open-label Clinical Study of Intratumoural Administration of BO-112 in Combination With Pembrolizumab in Subjects With Liver Metastasis From Colorectal Cancer or Gastric/Gastro-oesophageal Junction Cancer
Brief Title: Study of BO-112 With Pembrolizumab for Colorectal or Gastric/GEJ Cancer With Liver Metastasis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Highlight Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOT112-02; 2019-004624-38 (EudraCT Number); KEYNOTE-A06 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2020-08-05; First posted 2020-08-11 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer; Gastric Cancer; Oesophageal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Esophageal Neoplasms | interventions — BO-112; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Open-label, non-comparative study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Cohort A consisted of 11 patients with CRC (microsatellite stable [MSS]) with nonresectable liver metastases suitable for IT injection and who had received at least 2 prior standard of care systemic anticancer therapies for advanced/metastatic disease. Patients who had resection of hepatic metastases and had hepatic recurrence, needed to have 1 or more prior standard of care systemic anticancer therapies in order to be eligible for this study. BO-112 was administered in the liver metastasis at the dose of 1mg (1.2 mL) in combination with intravenous pembrolizumab given at the fixed dose of 200 mg, every 3 weeks for up to 35 cycles (2 years). During the first cycle, BO-112 was administered on D1 and D8.
  Interventions: Procedure: Hepatic Biopsy; Drug: BO-112 with pembrolizumab
- Cohort B (Experimental): Cohort B consisted of 7 patients with gastric or GC/GEJ with nonresectable liver metastases suitable for IT injection and who had received at least 1 prior standard of care systemic anticancer therapy for advanced/metastatic disease. BO-112 was administered in the liver metastasis at the dose of 1 mg (1.2 mL) in combination with intravenous pembrolizumab given at the fixed dose of 200 mg, every 3 weeks for up to 35 cycles (2 years). During the first cycle, BO-112 was administered on D1 and D8.
  Interventions: Procedure: Hepatic Biopsy; Drug: BO-112 with pembrolizumab

INTERVENTIONS:
Procedure: Hepatic Biopsy — In this trial a biopsy from the hepatic lesion to be injected will be mandatory on C1D1 and C2D1, prior to the BO-112 administration. On the same timepoints, a biopsy from a non-hepatic, non-injected lesion will be optional.
Drug: BO-112 with pembrolizumab — BO-112 was administered in the liver metastasis at the dose of 1mg (1.2 mL) in combination with intravenous pembrolizumab given at the fixed dose of 200 mg, every 3 weeks for up to 35 cycles (2 years). During the first cycle, BO-112 was administered on D1 and D8.
  Other Names: KEYTRUDA®

SUMMARY:
This is an open, single arm, multicenter phase 2 trial in which BO-112 will be administered intratumorally in combination with intravenous pembrolizumab in patients with liver metastasis from colorectal, gastric or gastroesophageal junction cancers. The objective is to reverse the primary resistance that a subgroup of patients from these tumors having microsatellite stability present to the PD-1 inhibitors. Treatment will be administered every 3 weeks, with the exception of the first cycle, in which BO-112 will be also administered on D8, for up to 2 years.

The primary objective is overall response rate based on RECIST 1.1 and safety, specifically referred to treatment emergent adverse events (TEAEs) with severity ≥ Grade 3 related to the study treatment (NCI-CTCAE v 5.0). The secondary endpoints include other efficacy endpoints (duration of response, disease control rate, progression-free survival, overall survival at 6 months, all based on RECIST 1.1, and overall response rate based on a specific tumor assessment criteria to evaluate the response to immunotherapies, IRECIST) and safety, in this case considering the number and proportion of subjects with treatment TEAEs (any grade) . In addition, the changes in the tumor microenvironment induced by the injection of BO-112 will be also evaluated as exploratory endpoints.

DETAILED DESCRIPTION:
The purpose of this Phase II study is to evaluate the safety, tolerability, antitumoural activity and systemic exposure of repeated IT administrations of BO-112 percutaneously injected into a hepatic metastatic lesion in combination with pembrolizumab administered intravenously.

This is an open-label, non-comparative, 2-cohort study with a Simon's 2-stage design which will include up to 69 evaluable adult subjects with un resectable liver metastasis suitable for IT injection from CRC or GC/GEJ who are naive to anti-PD1/PDL1 therapy.

Cohort A will consist of up to 26 subjects with metastatic CRC who have received at least 2 prior standard of care systemic anticancer therapies for advanced/metastatic disease. Bevacizumab may have been previously administrated. Prior Anti-EGFR drugs are mandatory if applicable depending on the RAS status.

Cohort B will consist of up to 43 subjects with gastric or GC/GEJ who have received at least 1 prior standard of care systemic anticancer therapy for advanced/metastatic disease. Prior Her2 blockade will be mandatory in those patients with Her2 positive tumors.

The aim of this study is to reverse the primary resistance that the subgroup of patients from these 2 cohorts who present microsatellite stability (MSS), in which data from previous clinical trials have demonstrate that the inhibition of PD-1 has no proven efficacy. For that purpose, the MSI status will be determined in the pre-treatment biopsy, done on C1D1, before the first BO-112 administration. Those patients with a MSI status will continue under study treatment but will be replaced and will not be considered for the efficacy assessment, only for the safety assessment. Those patients having a MSS status will be considered bot both assessments.

The recommended dose for further clinical development of BO-112 is 1 mg administered in 1.7 mL volume, based on the data from the 112/2016-IT study, the fist-in-human trial with BO-112. The planned dose of pembrolizumab for this study is 200 mg. Study treatment will consist of BO-112 IT injections in combination with IV pembrolizumab infusions and will be administered in 3-week cycles. For each cycle, BO-112 IT injections will be administered after the pembrolizumab infusion, either the same day or within a period of up to 36 hours after the pembrolizumab infusion (for organisational feasibility at the site). On the first cycle, BO-112 will be administered on D1 and D8.

The BO-112 IT injections will be administered by an interventional radiologist under ultrasound guidance, or occasional CT scan guidance, at the discretion of the interventional radiologist.

Study treatment should continue as long as there is clinical benefit and it is tolerated, up to a maximum of approx. 2 years (corresponding to 35 treatment cycles).

ELIGIBILITY:
Inclusion Criteria:

* Nonresectable liver metastasis(es) of colorectal or gastric/gastro-oesophageal junction cancer (GC/GEJ). History of resection for liver metastasis is allowed.
* Histological or cytological proof of colorectal (Cohort A) or GC/GEJ cancer (Cohort B).
* Progression during or after, or have not tolerated therapy for advanced/metastatic disease as follows:

  1. Cohort A (CRC): at least 2 lines of fluoropyrimidine, irinotecan and/or oxaliplatin containing therapy with or without bevacizumab; if epidermal growth factor receptor (EGFR) positive/RAS wild type, prior anti-EGFR treatment is required. Incase of prior resection of hepatic metastasis with hepatic recurrence, only 1 prior line of fluoropyrimidine, irinotecan and/or oxaliplatin containing therapy is required.
  2. Cohort B (GC/GEJ): fluoropyrimidine and platinum containing treatment; if Human epidermal growth factor receptor 2 (HER-2) positive, also prior anti-HER-2 treatment is required.
* At least 1 liver metastasis of minimum 20 mm in diameter that is suitable for percutaneous, IT injection .
* Presence of at least 1 measurable lesion according to RECIST v1.1. Note: this may be the liver metastasis selected for injection if it is the only measurable lesion present.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate haematologic and end-organ function

EXCLUSION CRITERIA

* Prior treatment with an anti-PD1, anti-PDL1 or anti-PDL2 agent, an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX40, CD137) or any Toll-like receptor (TLR) agonist.
* Liver metastasis(es) with macroscopic tumour infiltration into the main portal vein, hepatic vein or vena cava.
* Contraindications to tumour biopsy and injections of the hepatic metastasis(es).
* Chemotherapy, definitive (curative) radiation, or biological cancer therapy within 4 weeks prior to the first dose of study treatment.
* Palliative radiotherapy (≤ 2 weeks of radiotherapy) within 1 week of start of study treatment.
* Clinically active central nervous system (CNS) metastases and/or carcinomatosis meningitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanesa Pons, MD, PhD, Study Director — Highlight Therapeutics
Locations (12):
- Belgium (4):
  - Institut Jules Bordet, Brussels
  - UCL St-Luc, Brussels
  - University Hospital Antwerp (UZA), Edegem
  - Universitair Ziekenhus Gent, Ghent
- Italy (2):
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Azienda Ospedaliera Ospedale Niguarda Ca'Granda, Milan
- Spain (6):
  - Hospital Reina Sofía, Córdoba, Cordoba
  - Hospital Valle Hebrón, Barcelona
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Clínica Universitaria de Navarra, Pamplona
  - Hospital Clínico de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang X, Ge X, Zhang Y, Xue X. The current management and biomarkers of immunotherapy in advanced gastric cancer. Medicine (Baltimore). 2022 May 27;101(21):e29304. doi: 10.1097/MD.0000000000029304. PMID 35623069
- See also: Company web site — http://www.highlighttherapeutics.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Cohort A consisted of 11 patients with CRC (microsatellite stable [MSS]) with nonresectable liver metastases suitable for IT injection and who had received at least 2 prior standard of care systemic anticancer therapies for advanced/metastatic disease. Patients who had resection of hepatic metastases and had hepatic recurrence, needed to have 1 or more prior standard of care systemic anticancer therapies in order to be eligible for this study.
- Cohort B: Cohort B consisted of 7 patients with gastric or GC/GEJ with nonresectable liver metastases suitable for IT injection and who had received at least 1 prior standard of care systemic anticancer therapy for advanced/metastatic disease.
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 11 | 7
Completed | 0 | 0
Not Completed | 11 | 7
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — progressive disease | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 11 | 7 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 11
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Full Range); unit: years] | 55.6 [37 to 74] | 56.1 [37 to 71] | 55.8 [37 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 7 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 1 | 1 | 2
  Italy | 1 | 0 | 1
  Spain | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Anti-tumour Efficacy:Overall Response Rate (ORR) Based on RECIST 1.1
Description: ORR based on the best objective response (BOR) using RECIST 1.1 of repeated IT administrations of BO-112 in metastatic liver lesions in combination with IV pembrolizumab
Time Frame: from baseline to approximately 8 months
Population: Cohort B: only 5 patients were evaluable for efficacy with one baseline and at least one on treatment efficacy assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort B: Cohort B consisted of 7 patients with gastric or GC/GEJ with nonresectable liver metastases suitable for IT injection and who had received at least 1 prior standard of care systemic anticancer therapy for advanced/metastatic disease. Only 5 patients were evaluable for efficacy with baseline and at least one on treatment efficacy assessment. BO-112 was administered in the liver metastasis at the dose of 1 mg (1.2 mL) in combination with intravenous pembrolizumab given at the fixed dose of 200 mg, every 3 weeks for up to 35 cycles (2 years). During the first cycle, BO-112 was administered on D1 and D8.
  Hepatic Biopsy: In this trial a biopsy from the hepatic lesion to be injected will be mandatory on C1D1 and C2D1, prior to the BO-112 administration. On the same timepoints, a biopsy from a non-hepatic, non-injected lesion will be optional.
  BO-112 with pembrolizumab: BO-112 was administered in the liver metastasis at the dose of 1mg (1.2 mL) in combination with intravenous pembrolizumab given at the fixed dose of 200 mg, every 3 weeks for up to 35 cycles (2 years). During the first cycle, BO-112 was administered on D1 and D8.
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 5
Participants | 0 | 0

2. Primary Outcome: Safety: Adverse Events
Description: Number and proportion of subjects with study treatment-related TEAEs with severity Grade 3 and higher (NCI-CTCAE v 5.0)
Time Frame: from baseline to approximately 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 7
Participants | 4 | 4

3. Secondary Outcome: Disease Control Rate Based on RECIST 1.1
Description: Best response for CR, PR as well as stable disease (SD) using RECIST 1.1
Time Frame: from baseline to approximately 8 months
Population: Cohort B: only 5 patients were valid for efficacy with one baseline and at least one on-treatment efficacy assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 5
Participants | 0 | 0

4. Secondary Outcome: Objective Response Rate Based iRECIST
Description: Based on best overall response using RECIST modified for immune-based therapies (iRECIST)
Time Frame: from baseline to approximately 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 5
Participants | 0 | 0

5. Secondary Outcome: Disease Control Rate Based on iRECIST
Description: Comprising best response for CR, PR as well as SD using iRECIST
Time Frame: from baseline to approximately 8 months
Population: Cohort B: only 5 patients were evaluable for efficacy with one baseline and at least one on-treatment efficacy assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 5
Participants | 0 | 0

6. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS)
Time Frame: from baseline to approximately 8 months
Population: Cohort B: only 5 patients were evaluable for efficacy with one baseline and at least one on-treatment assessment
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 5
months | 1.35 [1.02 to 1.41] | 1.38 [0.95 to 2.56]

7. Secondary Outcome: Overall Survival Rate
Description: Number of subjects alive at 6 months
Time Frame: at 6 months from enrolment
Population: only 5 patients were evaluable for efficacy with both baseline and at least one post-baseline imaging
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 5
Participants | 9 | 3

ADVERSE EVENTS:
Time Frame: from baseline to approximately 8 months
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 2/11 | 2/7
Serious Adverse Events (participants affected / at risk) | 5/11 | 2/7
Other Adverse Events (participants affected / at risk) | 11/11 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=11) | Cohort B (N=7)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
pyrexia (Gastrointestinal disorders) | 3 (3) | 0 (0)
alpha hemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
COVID 19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
bacteriemia (Infections and infestations) | 0 (0) | 1 (1)
syncope (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=11) | Cohort B (N=7)
pyrexia (General disorders) | 8 (20) | 4 (8)
Hypertension (Vascular disorders) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 3 (6) | 2 (2)
Chills (General disorders) | 5 (9) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (2)
Injection site pain (General disorders) | 0 (0) | 2 (5)
Cytokine release syndrome (Immune system disorders) | 2 (4) | 1 (3)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Eczema eyelids (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (12) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (7) | 2 (3)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Disuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Asymptomatic COVID-19 (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/40/NCT04508140/Prot_SAP_000.pdf